CLINICAL TRIAL: NCT03938623
Title: Teaching General Practitioners to Use the Patient-centered Approach When Suggesting Colorectal Cancer Screening
Acronym: FORCEPS
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Collège de la Médecine Générale, France (Other)
Collaborators: National Cancer Institute, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2016IAN913
Record Dates: First submitted 2019-04-25; First posted 2019-05-06 (Actual); Last update posted 2019-05-06 (Actual); Status verified 2019-04

CONDITIONS: Colorectal Cancer
Keywords: colorectal cancer; general practitioners; the patient-centered approach
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Training: Teaching general practitioners to use the patient-centered approach when suggesting colorectal cancer screening
  Interventions: Other: Training
- Control: General Practitioners not using the patient-centered approach

INTERVENTIONS:
Other: Training — Teaching general practitioners to use the patient-centered approach when suggesting colorectal cancer screening
  Other Names: The patient-centered approach
  Groups: Training

SUMMARY:
Context : Colorectal cancer (CRC) mass screening has been implemented in France since 2008. Participation rates remain too low. The objective of this study is to test if the implementation of a training course focused on communication skills (whether in-person or e-learning) among general practitioners (GP) would increase the delivery of gFOBT and CRC screening participation among the target population of each participating GP.

Method : Pragmatic controlled cluster randomized trial with 2 parallel groups: Control versus Educational Intervention Intervention ; six hour educational training either in person or through e-learning The Main objective: is to evaluate the effectiveness of an educational intervention teaching physicians the patient-centered approach, either in-person or through e-learning, by evaluating their patients' participation in colorectal cancer (CRC) screening for all risk categories.

DETAILED DESCRIPTION:
Context : Colorectal cancer (CRC) mass screening has been implemented in France since 2008. Participation rates remain too low. The objective of this study is to test if the implementation of a training course focused on communication skills (whether in-person or e-learning) among general practitioners (GP) would increase the delivery of gFOBT and CRC screening participation among the target population of each participating GP.

Method : Pragmatic controlled cluster randomized trial with 2 parallel groups: Control versus Educational Intervention .Given that the type of educational intervention modifies the global organization and medical practices of the participating centers, the randomization will be done at the level of GP's practice as a cluster unit in order to avoid contamination bias.

Population : All general practitioners practicing in the Île-de-France, Languedoc-Roussillon, Loire-Atlantique, Midi-Pyrénées, Poitou-Charentes, or Provence-Alpes-Cote-d'Azur regions will be requested Their patients are eligible if they are 50-74 years old and reside in one of the above regions.

212 centers are expected with 318 investigating doctors (an average of 1,5 doctors per center) and 42 358 total patients (21 179 patients in each arm) Intervention ; will be an educational training either in person or through e-learning GPs from practices in the control group were asked to continue their usual care, as if they were not participating in this trial. The whole procedure is the same all over the country i.e. all adults aged 50 to 74 of each GP's target population receive a letter every two years from the local cancer prevention association encouraging them to visit their GP and ask for the test. Patients must then send the test and a completed identity form, contained in an envelope to a central laboratory.

In the intervention group, participating GPs will receive a six-hour training course focusing on patient-centered care either in person or through e-learning . Two different scenarios for a video aiming to improve communication with patients were developed: one for a compliant patient, another for a non-compliant patient based on the four components of the patient centered clinical method

Objectives :

The Main objective: is to evaluate the effectiveness of an educational intervention teaching physicians the patient-centered approach, either in-person or through e-learning, by evaluating their patients' participation in colorectal cancer (CRC) screening for all risk categories The Secondary objectives are ;

* Assess the effectiveness of this training on moderate-risk patient participation in organized CRC screening
* Assess the effectiveness of this training on high-risk patient participation in targeted CRC screening
* Compare the effectiveness of in-person training versus e-learning
* Assess the effect of the training on whether the sequence of tests completed by patients is appropriate for their risk category (carrying out a test that was given to them, immediate refusal of the test, carrying out a colonoscopy if the test is positive) Assess the effectiveness of this training on reducing social inequalities in CRC screening participation Evaluation criteria : the primary endpoint is patient participation in the appropriate CRC screening for their level of risk (i.e. completing the Fecal Occult Blood Test [FOBT] if at moderate risk or a colonoscopy if at high risk) within 12 months of randomization. The secondary endpoints are: completing the FOBT for moderate risk patients, completing a colonoscopy for higher risk patients, proportion of dispensed tests that were completed , proportion of tests refused among those proposed, proportion of colonoscopies performed among those whose FOBT is positive, patient screening participation rate according to socio-economic level, proportion of tests that could not be interpreted

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 50 to 74,
* Residing in the regions of Île-de-France, Languedoc-Roussillon, Loire-Atlantique, Midi-Pyrenees, Poitou-Charentes, and Provence-Alpes-Côte-D'azur,
* Registered on the AMELI file of general practitioners participating in beginning of the study, before the training (ie the patients who have declared as a doctor one of the participating general practitioners).
* Affiliation to the general social security scheme

Exclusion Criteria:

* Patients excluded from screening for medical reasons (colorectal cancer or symptoms such as presence of red or black blood in the stool, other pathologies in non-priority treatment and screening)
* Patient having performed a Hemoccult® test / test immunological test for less than 2 years or had colonoscopy for less than 5 years.
* Patient who has declared as a treating physician one of the participating physicians for the duration of the study.
* Patient who did not consult for the duration of the study

Ages: 50 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All general practitioners practicing in the Île-de-France, Languedoc-Roussillon, Loire-Atlantique, Midi-Pyrénées, Poitou-Charentes, or Provence-Alpes-Cote-d'Azur regions will be requested Their patients are eligible if they are 50-74 years old and reside in one of the above regions.
Sampling Method: Probability Sample
Enrollment: 274 (Actual)
Dates: Start 2018-01-24 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
number of patients screened positive using the patient-centered approach after training of face to face training or e-learning | 1 year
  Evaluate the effectiveness of face to face training or e-learning training to use the patient-centered approach

CONTACTS AND LOCATIONS:
Overall Officials: AUBIN-AUGER M ISABELLE, MD, Pr, Principal Investigator — COLLEGE DE LA MEDECINE GENERALE
Locations (1):
- Département de Médecine Générale, Paris, Idf, France

IPD SHARING:
Plan to Share IPD: Undecided